CLINICAL TRIAL: NCT01406821
Title: Randomized, Double-blind Clinical Trial of Platelet Rich Plasma for Treatment of Acute and Chronic Patellar Tendinosis
Brief Title: Treatment of Acute and Chronic Ligament and Tendon Injuries With Platelet Rich Plasma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: NYU Langone Health (Other)
Responsible Party: Principal Investigator, Jason L. Dragoo, Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SU-10162010-7109; 16595
Record Dates: First submitted 2011-07-28; First posted 2011-08-01 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Tendinopathy
Keywords: PRP; platelet-rich-plasma; platelet; tendinosis; tendinitis; tendonitis; tendinopathy; enthesopathy; muscle; sport; tendon; patella; patellar tendon
MeSH Terms: conditions — Tendinopathy; Enthesopathy; Patella Fracture | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Dry needling (Sham Comparator): Blood will be drawn, and tendon will be penetrated with dry needle. Nothing will be injected into the tendon.
  Interventions: Procedure: Ultrasound-guided dry needling
- Platelet-rich plasma (PRP) (Experimental): Blood will be drawn, and platelet-rich plasma will be injected into the tendon.
  Interventions: Procedure: Ultrasound-guided platelet-rich-plasma (PRP) injection

INTERVENTIONS:
Procedure: Ultrasound-guided platelet-rich-plasma (PRP) injection — Blood will be drawn, and platelet-rich plasma will be injected into the tendon under ultrasound guidance.
  Arms: Platelet-rich plasma (PRP)
Procedure: Ultrasound-guided dry needling — Blood will be drawn, and tendon will be penetrated with dry needle under ultrasound guidance. Nothing will be injected into the tendon.
  Arms: Dry needling

SUMMARY:
Platelet rich plasma has been used in previous studies to stimulate faster healing of torn ligaments and tendons in order to help reduce pain and restore normal function. This study aims to prove that non-operative treatment of acute and chronic ligament and tendon injuries with platelet rich plasma will reduce the time needed for participants to heal these injuries and restore function.

We are currently enrolling patients with PATELLAR TENDON INJURIES in the KNEE.

DETAILED DESCRIPTION:
Pre-procedure diagnosis: The appropriate clinical evaluation will be dictated by the examining physician. Minimal pre-procedure studies will include plain radiographs and MRI. All patients will complete a pretreatment questionnaire.

Patients will be randomized and blinded to a treatment regimen.

Method of randomization: Some of the participating subjects will receive platelet rich plasma and others will receive a saline injection. The platelet rich plasma experimental group will have up to 50cc of whole blood collected via venipuncture and prepared using the standard PRP protocol.

To blind the control group these patients will have a simulated needle stick and approximately 10 ml (2 teaspoons) of blood will be drawn. No blood will be given back to the patient. For those in the control group their ligament or tendon will be stimulated with dry needling (moving a needle up and down in the tendon, without injection). Patients in the PRP treatment group will also have dry needling, plus the PRP will be injected into the tendon as well.

Platelet rich plasma injections have an equivalent risk profile to routine injections. Those potential risks include skin discoloration, pain at injection site, superficial or deep infection, no relief of symptoms, worsening of symptoms, and damage to nerve and blood vessels. Potential benefits include significant improvement in symptoms and reduction in time for return to function.

Post injection activity: All patients will use crutches for 24-48 hours after injection. All patients will have physical therapy two times a week according to a standardized protocol.

Follow up at the clinic for all patients will be every 3 weeks from weeks 1-12. All patients will fill out an injury location specific questionnaire, Tegner Activity Scale, short form-12, and visual analog scale for pain, among others. Additional follow-up will be done at 6 months, 1 year and 2 years. All radiographic studies will be read by a radiologist blinded to the study groups.

The primary endpoint for all patients in the study will be twelve weeks. Secondary enpoints are 6 months, 1 year and 2 years.

ELIGIBILITY:
Inclusion Criteria:

-Acute or chronic ligament or tendon injuries

Exclusion Criteria:

* Pregnant women,
* children,
* other injuries that require surgical intervention,
* associated fractures,
* systemic disease resulting in an immunocompromised state affecting ability to heal soft tissues

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-08 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Patient-reported improvement in symptoms at 12 weeks | 12 weeks

SECONDARY OUTCOMES:
Reduction in patellar tendinosis by MRI | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Christina Herrero, Study Director — New York University Langone Orthopedic Hospital; Dr. Jason L. Dragoo, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Stanford University School of Medicine, Stanford, California
  - New York University Langone Orthopedic Hospital, New York, New York

IPD SHARING:
Plan to Share IPD: No